CLINICAL TRIAL: NCT05189275
Title: Cannabidiol and Focus Study (CBD-Focus)
Acronym: CBD-Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28497
Record Dates: First submitted 2021-11-20; First posted 2022-01-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Cannabidiol

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to 1 of 4 groups and followed throughout the 8 week intervention period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cannabidiol 40 mg (CBD40) (Experimental): Subjects consume beverages with 40mg of CBD.
  Interventions: Dietary Supplement: Daily Beverage Intervention
- Cannabidiol 20 mg (CBD20) (Experimental): Subjects consume beverages with 20mg of CBD.
  Interventions: Dietary Supplement: Daily Beverage Intervention
- Cannabidiol 0 mg (CBD0) (Experimental): Subjects consume beverages with 0mg of CBD.
  Interventions: Dietary Supplement: Daily Beverage Intervention
- Placebo Beverage (PLAC) (Placebo Comparator): Subjects consume calorie matched beverages with 0 CBD.
  Interventions: Dietary Supplement: Daily Beverage Intervention

INTERVENTIONS:
Dietary Supplement: Daily Beverage Intervention — Individuals will consume one of 4 beverages, daily for 8 weeks.

SUMMARY:
Cannabidiol (CBD), a non-psychoactive hemp derivative, is an attractive therapeutic target, and is most supported by the scientific community as an antiepileptic, anxiolytic, and antipsychotic. Additionally, CBD may cause alterations in aspects of health and fitness, fatigue, stress, calmness, quality of life, cognitive function, ability to maintain focus, sleep quantity, and sleep quality. Cannabidiol may be associated with alterations in inflammatory response in the human body, which has implications in both healthy and diseased populations. Natural killers cells (NKC) play a vital role in maintain your body's defenses and are an essential component of your immune system. In humans, NKC contain the highest concentrations of receptors associated with the endocannabinoid system and CBD. Human models have demonstrated that CBD use increases the percentage of NKC in peripheral blood. However, similar models found that CBD administration inhibits markers of NKC cytotoxic function, a beneficial cellular mechanism used to prevent malignant cell transformation and viral infection. The overarching goal of this investigation is to determine the effects of an 8-week CBD intervention on measures of fatigue, stress, calmness, quality of life, cognitive function, focus, health and fitness, and sleep quantity, and sleep quality. In addition, this study will explore a potential CBD mechanism of action with a focus on biomarkers of neural health, inflammation, liver health, kidney health, as well as NKC number and function.

DETAILED DESCRIPTION:
BACKGROUND: Cannabidiol (CBD), a non-psychoactive hemp derivative, is an attractive therapeutic target, and is most supported by the scientific community as an antiepileptic, anxiolytic, and antipsychotic. Additionally, CBD may cause alterations in aspects of health and fitness, fatigue, stress, calmness, quality of life, cognitive function, ability to maintain focus, sleep quantity, and sleep quality. Cannabidiol may be associated with alterations in inflammatory response in the human body, which has implications in both healthy and diseased populations. In humans, natural killer cells (NKC) contain the highest concentrations of receptors associated with the endocannabinoid system and CBD. Human models have demonstrated that CBD use increases the percentage of NKC in peripheral blood. However, similar models found that CBD administration inhibits markers of NKC cytotoxic function, a beneficial cellular mechanism used to prevent malignant cell transformation and viral infection. The overarching goal of this investigation is to determine the effects of an 8-week CBD intervention on measures of fatigue, stress, calmness, quality of life, cognitive function, focus, health and fitness, and sleep quantity, and sleep quality. In addition, this study will explore a potential CBD mechanism of action with a focus on biomarkers of neural health, inflammation, liver health, kidney health, as well as NKC number and function.

METHODS: In this double-blind, placebo-controlled, 4 arm clinical trial, male and female participants will undergo 2 pre intervention study visits and 3 post intervention study visits separated by an 8-week intervention period. Participants must be aged 18-50 years old, currently completing at least 150 minutes of moderate to vigorous physical activity per week, have a body mass index under 29.9, with no significant physical or mental health (without the presence of chronic depression or anxiety) conditions. Subjects may not have an allergy to soy. All study subjects must also be free of cannabis product use or regular high doses of antioxidants for the previous 8 weeks. Supplementation groups will be randomly assigned into groups consuming one of 4 beverages: 1) a beverage with 40 mg of CBD (CBD40, n=50), 2) a beverage with 20 mg of CBD (CBD20, n=50), 3) a beverage with 0 mg of CBD (CBD0, n=50) or 4) calorie-matched placebo (PLAC, n=50).

INTERVENTION DESCRIPTION: Participants will be instructed to consume one beverage per day following their last meal, 1-1.5h before bed. Four weeks of beverages will be provided at a time. These beverage deposits will include an in person check in at the midpoint of the study. Participants and researchers will be blinded to the intervention groups. All participants will be given a 4-week supply of beverages. Investigators will meet with participants weekly via zoom/phone call and to report any adverse side effects or changes in physical activity routine. All products will be provided by Ocean Spray. All products are hemp derived, within legal limits and have had their purity verified. Following the completion of data collection for all study participants, researchers will be unblinded to supplementation groups.

ELIGIBILITY:
Inclusion Criteria:

* Currently completing at least 150 minutes of moderate to vigorous physical activity per week
* Have a body mass index under 29.9
* No significant physical or mental health (without the presence of chronic depression or anxiety) conditions
* No presence or past diagnosis of eating disorders

Exclusion Criteria:

* Subjects may not have an allergy to soy.
* All study subjects must also be free of cannabis product use or regular high doses of antioxidants for the previous 8 weeks.

Participants receive a $200 Visa Gift Card after the last study visit is completed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life Questionnaire Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Ferrans and Powers Quality of Life Index Questionnaire. A higher scores suggests higher quality of life.
Change in Fatigue Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Piper Fatigue Questionnaire. A higher score suggests higher levels of fatigue.
Change in Sleep Assessment | Just before the 8 Week Intervention and in the 7th Week of the 8 Week Intervention
  Sleep Assessment (7 day). We will use Fitbits to track sleep.
Change in Sleep Questionnaire Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Leeds Sleep Questionnaire. Lower scores generally suggest better sleep.
Change in Physical Activity (steps per day) | Just before the 8 Week Intervention and in the 7th Week of the 8 Week Intervention
  Physical Activity Assessment (7 day). We will use Fitbits to track physical activity.
Change in Perceived Stress Scale Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Perceived Stress Questionnaire. A higher score suggests higher perceived stress.
Change in General Anxiety Disorder Questionnaire Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  General Anxiety Disorder Questionnaire 7. A higher score suggests higher levels of anxiety.
Change in Psychological Wellbeing Scale Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Psychological Wellbeing Questionnaire. A higher score suggests better wellbeing.
Change in Cognitive Function and Abilities Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function Abilities - Short Form 8a. A higher score suggests higher cognitive ability.
Change In Cognitive Function Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  PROMIS Cognitive Function - Short Form 8a. A higher score suggests higher cognitive ability.
Change in Athlete Sickness and Illness Assessment Score | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  The Wisconsin Upper Respiratory Symptom Survey. A higher scores suggests more respiratory symptoms.
Change in Sustained Attention to Response Task (SART) Activity | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Sustained Attention to Response Task (SART) Activity
Change in Maximal Anaerobic Power | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Wingate Power Test
Change in Natural Killer (NK) Cell Number | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  NK Cell Counts obtained on a flow cytometer.
Change in Natural Killer (NK) Cell Function | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  NK Cell Cellular Function Assay using Flow Cytometry
Change in a Biomarker of Inflammation | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Serum C-Reactive Protein
Change in a Biomarker of Neural Health | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Circulating Brain Derived Neurotropic Factor
Change in a Stress Biomarker | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Serum Cortisol
Change in Liver Health Biomarker I | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Serum Aspartate aminotransferase (AST)
Change in Liver Health Biomarker II | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Serum Alanine aminotransferase (ALT)
Change in Kidney Health Biomarker | Just before the 8 Week Intervention and Immediately Following the 8 Week Intervention
  Serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: James Haughian, PhD, Principal Investigator — University of Northern Colorado; Laura K Stewart, PhD, Principal Investigator — University of Northern Colorado
Locations (1):
- University Of Northern Colorado, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will become available when the study is published and will be available for 3 years.
Supporting Information: Study Protocol
Time Frame: Data will become available when the study is published and will be available for 3 years.
Access Criteria: Data (without subject ID numbers) will be shared upon email request laura.stewart@unco.edu.